CLINICAL TRIAL: NCT00034450
Title: Developmental Study on Fatigue in Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: R21AT001025-01 (NIH); NCT00060034 (obsolete NCT alias)
Record Dates: First submitted 2002-04-29; First posted 2002-04-30 (Estimated); Last update posted 2006-08-18 (Estimated); Status verified 2006-03

CONDITIONS: Neoplasms
Keywords: Terminal Cancer
MeSH Terms: conditions — Neoplasms | interventions — Carnitine

INTERVENTIONS:
Drug: L-carnitine

SUMMARY:
L-carnitine is a supplement (type of vitamin) that has been suggested to be decreased in patients with cancer. We will identify patients that have terminal cancer and fatigue. The purpose of this study is to determine if L-carnitine replacement improves fatigue in cancer patients with L-carnitine deficiency.

DETAILED DESCRIPTION:
Fatigue is the most frequently reported symptom in patients with cancer. The causes of fatigue are multifactorial and include the disease itself, antineoplastic therapies, anemia, depression, and malnutrition. Our preliminary data suggest that micronutrient deficiencies, specifically carnitine deficiency, may be an important factor in fatigue. Carnitine plays a major role in energy metabolism. Systemic depletion is characterized by weight loss, fatigue, muscle weakness, decreased tolerance to metabolic stress, and cardiomyopathy. We found deficiency of the micronutrient carnitine in 17/27 patients with cancer. Symptoms of fatigue and functional status improved significantly in those patients who received oral L-carnitine supplementation. In addition, we observed similar results in 6/10 patients with end stage AIDS presenting with carnitine deficiency. Objectives: a) To determine the effect of L-carnitine therapy on symptoms of fatigue in patients with terminal cancer and serum carnitine deficiency, and b) to determine the effect of L-carnitine therapy on performance status, cognitive function, mood, quality of life, and motor activity in these patients. Study Design: We propose to conduct a Phase Il developmental randomized double-blind placebo-controlled study to determine the effect of the micronutrient L-carnitine on fatigue and other outcomes in patients with terminal cancer. A sample of 130 patients with terminal cancer, fatigue and serum carnitine deficiency will be recruited into the intervention study. At the first visit, the patients will receive a baseline assessment of fatigue, performance status, cognitive function, mood, and quality of life and motor activity. a) During weeks 1-4, patients will be randomized to receive L-carnitine, 2 g/day, placebo. b) During weeks 5-8, all patients will receive L-carnitine at a dose of 2 g/day, for a period of 4 weeks. Measures will be repeated at 48 hs, 2 weeks, 4 weeks and 8 weeks. The primary endpoint will be change in fatigue at 4 weeks. Analysis will evaluate group differences in the primary endpoint and other outcomes. An interim analysis will be done once 15 patients have been observed in each group at 4 weeks. Paired and unpaired data analyses between groups will be conducted with the assistance of a statistician.

ELIGIBILITY:
Inclusion:

* Patients with diagnosis of cancer and estimated life expectancy of less than 6 months.
* Patients who have undergone antineoplastic therapy which may worsen fatigue or promote carnitine deficiency will be eligible if completed the therapy more than 90 days prior to beginning the study.

Exclusion:

* Uncontrolled or severe cardiovascular, pulmonary, or renal disease.
* Patients with encephalopathy or psychiatric disorder sufficiently severe to impair completion of the questionnaire.
* Treatment or replacement therapy with any form of carnitine less than 12 months prior to enrollment.
* Known sensitivity to carnitine.
* History of seizures or stroke.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140
Dates: Start 2002-01; Study Completion 2004-08

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo A. Cruciani, MD, PhD, Principal Investigator — Beth Israel Medical Center, Department of Pain Medicine and Palliative Care
Locations (1):
- Beth Israel Medical Center, New York, New York, United States